CLINICAL TRIAL: NCT05343429
Title: ''Comparison of Preoperative Aspirin and Benzydamine Hydrochloride Gargles on Reduction in Severity and Duration of Post-Operative Sore Throat. A Randomized Controlled Parallel Study.''
Brief Title: Preoperative Aspirin and Benzydamine Hydrochloride Gargles on Severity and Duration of Post-Operative Sore Throat
Acronym: Postbenas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Mohammad Shafiq, Consultant Anesthesiologist, Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RMI/RMI-REC/Approval/122
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Benzydamine; Long-Term Synaptic Depression; Aspirin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment The study design is prospective double-blinded randomized controlled parallel trial with allocation ratio of 1:1.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: A pharmacist not part of the study will prepare two solutions, one of Benzydamine hydrochloride (BH) 0.15 % 15 ml diluted to 30 ml by adding plain water and another of Aspirin (AS) 600 mg dissolved in 30 ml plain water. The randomized patients will gargle with either BH and AS solution five minutes before conduct of General Anesthesia. The unique identification will be known only to principal investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benzydamine hydrochloride (BN) (Active Comparator): 15 ml of 0.15 % Benzydamine hydrochloride (BN) to dissolved in 15 ml plain water in a sterile container
  Interventions: Drug: Benzydamine hydrochloride
- Aspirin (Ap) (Active Comparator): 600 mg Aspirin tablets dissolved in 30 ml of plain water
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Benzydamine hydrochloride — In BN group,15 ml of 0.15 % Benzydamine hydrochloride (BN) will be dissolved in 15 ml plain water in a sterile container and given to participants before anesthesia for surgery
  Other Names: BENZIRIN oral rinse 240ml by Adamjee Pharmaceuticals (Pvt.) Ltd.
  Arms: Benzydamine hydrochloride (BN)
Drug: Aspirin — In group AP, Aspirin (AP) 600 mg Aspirin tablets dissolved in 30 ml of plain water in a sterile container will be given to participants for gargling before anesthesia for surgery
  Other Names: Tablets. Disprin 300 mg (soluble) by by Reckitt Benckiser (Pvt.) Ltd.
  Arms: Aspirin (Ap)

SUMMARY:
Post-operative sore throat (POST) following General Anesthesia with endotracheal is a common symptom and drains resources. The researchers will compare preoperative gargling of Asprine and Benzydamine HCL to study comparative effects on intensity and duration of POST. Data collected as such will be analyzed to reach at a conclusion.

DETAILED DESCRIPTION:
Endotracheal intubation commonly causes postoperative sore throat (POST). Its incidence is 22 - 62% in the adult population whereas in children the incidence is 24 to 44%. In adult population peak incidence is 2 to 4 hours after tracheal extubation. There is a limited medical literature available about incidence and peak time of occurrence after tracheal extubation in children. Though relieved in due course of time, POST leads to postoperative dissatisfaction. Traumatic laryngoscopy and endotracheal tube residence are the most likely offenders individually or combined. Other risk factors include preexisting upper respiratory tract infection, multiple intubation attempts, intubating un-paralyzed patient, high ETT cuff pressure, prolonged anesthesia with ETT and inexperienced operator.

The problem i.e. POST preemptive amelioration, has been studied using various pharmacological interventions. The list includes, but is not limited to, Benzydamine hydrochloride, aspirin, ketamine, lidocaine and dexamethasone. In a study conducted by Agarwal A, Nath SS, Goswami D et al on adult female patients employing preoperative Aspirin and Benzydamine hydrochloride gargling found it simple, safe and effective method in reducing incidence and severity of POST. Their patients were scheduled for mastectomy. However, a study conducted by Hyung-Been Yhim, Soo-Hyuk Yoon, Young-Eun Jang et al in pediatrics was unsuccessful to show reduction in POST when they used Benzydamine hydrochloride (BH) spray on vocal cords and upper airway before tracheal intubation. They asked for more research and suggested well-designed and powered RCT's in children. The current study will differ from previously conducted research and will include adult males of different ethnicity and type of surgery.

Objectives: To compare the effect of Aspirin and Benzydamine hydrochloride (BH) gargles on incidence, severity and duration of POST.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists Class 1 and 2 (ASA 1 and 2) scheduled for gynecological surgery under General Anesthesia with Intra tracheal Intubation and expected to finish in less than three hours will be included in the study.
* Patients of 18- 60 years of age will be included.
* Patients of Mallampati class 1 and 2 will be selected, as these have easy intubation predicted.
* Patients qualifying for easy intubation (prediction based on mouth opening, neck mobility etc.) will be selected.
* Patients in supine position only.

Exclusion Criteria:

* Patients who are unable to gargle properly.
* Patients who require more than 2 attempts at intubation.
* Patients of Cormack-Lehane Grade 3 and 4 on direct laryngoscopy (multiple intubating attempts may be required).
* Patients requiring oral cavity instrumentation e.g. N/G tube placement, oral or laryngeal surgeries including tonsillectomies
* Patients whose head are frequently turned > 90 degrees with ETT placed in.
* Patients whose surgery is prolonged beyond 3 hour.
* Patients who require postoperative mechanical ventilation.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative sore throat (POST) in both groups | Six hours
  Rate (incidence) of Postoperative sore throat (POST) in both groups will be calculated and compared with each other.

SECONDARY OUTCOMES:
Duration of Postoperative sore throat (POST) in both groups | Six hours post-operative period
  Based on structured proforma, participants will be followed for any complaints of POST at regular intervals and duration of POST will be calculated and compared.
Severity of Postoperative sore throat (POST) in both groups | Six hours post-operative period
  Severity of Postoperative sore throat (POST) in both groups will be assessed and compared. POST will be graded on a 4-point scale i.e. 0 through 3. 0 for no sore throat, 1 for mild sore throat (complaints of sore throat only upon asking), 2 for moderate sore throat (complaints of sore throat at one's own), and 3 for severe sore throat (change of voice / hoarseness; and associated with throat pain).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Shafiq, FCPS, Principal Investigator — Rehman Medical institute, Pakistan
Locations (1):
- Rehman Medical Institute, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Yes Data including clinical and demographic characteristics, not affecting patient's confidentiality, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April, 2022 to April, 2025
Access Criteria: IPD will be shared on inter institutional request basis.

REFERENCES:
- [Background] Chandler M. Tracheal intubation and sore throat: a mechanical explanation. Anaesthesia. 2002 Feb;57(2):155-61. doi: 10.1046/j.1365-2044.2002.02329.x. PMID 11871952
- [Result] Piriyapatsom A, Dej-Arkom S, Chinachoti T, Rakkarnngan J, Srishewachart P. Postoperative sore throat: incidence, risk factors, and outcome. J Med Assoc Thai. 2013 Aug;96(8):936-42. PMID 23991600
- [Result] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Result] Calder A, Hegarty M, Erb TO, von Ungern-Sternberg BS. Predictors of postoperative sore throat in intubated children. Paediatr Anaesth. 2012 Mar;22(3):239-43. doi: 10.1111/j.1460-9592.2011.03727.x. Epub 2011 Nov 8. PMID 22066487
- [Result] Patki A. Laryngeal mask airway vs the endotracheal tube in paediatric airway management: A meta-analysis of prospective randomised controlled trials. Indian J Anaesth. 2011 Sep;55(5):537-41. doi: 10.4103/0019-5049.89900. PMID 22174478
- [Result] Mostafa RH, Saleh AN, Hussein MM. A comparative study of three nebulized medications for the prevention of postoperative sore throat in the pediatric population. Open Anesthesia J. 2018;12(1):85-93.
- [Result] Chen CY, Kuo CJ, Lee YW, Lam F, Tam KW. Benzydamine hydrochloride on postoperative sore throat: a meta-analysis of randomized controlled trials. Can J Anaesth. 2014 Mar;61(3):220-8. doi: 10.1007/s12630-013-0080-y. Epub 2013 Nov 22. PMID 24263969
- [Result] Agarwal A, Nath SS, Goswami D, Gupta D, Dhiraaj S, Singh PK. An evaluation of the efficacy of aspirin and benzydamine hydrochloride gargle for attenuating postoperative sore throat: a prospective, randomized, single-blind study. Anesth Analg. 2006 Oct;103(4):1001-3. doi: 10.1213/01.ane.0000231637.28427.00. PMID 17000820
- [Result] Mayhood J, Cress K. Effectiveness of ketamine gargle in reducing postoperative sore throat in patients undergoing airway instrumentation: a systematic review. JBI Database System Rev Implement Rep. 2015 Sep;13(9):244-78. doi: 10.11124/jbisrir-2015-2045. PMID 26470672
- [Result] Tanaka Y, Nakayama T, Nishimori M, Tsujimura Y, Kawaguchi M, Sato Y. Lidocaine for preventing postoperative sore throat. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD004081. doi: 10.1002/14651858.CD004081.pub3. PMID 26171894
- [Result] Kuriyama A, Maeda H. Preoperative intravenous dexamethasone prevents tracheal intubation-related sore throat in adult surgical patients: a systematic review and meta-analysis. Can J Anaesth. 2019 May;66(5):562-575. doi: 10.1007/s12630-018-01288-2. Epub 2019 Jan 7. PMID 30617677
- [Result] Yhim HB, Yoon SH, Jang YE, Lee JH, Kim EH, Kim JT, Kim HS. Effects of benzydamine hydrochloride on postoperative sore throat after extubation in children: a randomized controlled trial. BMC Anesthesiol. 2020 Apr 4;20(1):77. doi: 10.1186/s12871-020-00995-y. PMID 32247315